CLINICAL TRIAL: NCT02045810
Title: Surgical Pleth Index - Relevance in Small Children. A Randomised Double Blinded Study
Brief Title: Surgical Pleth Index- Relevance in Small Children
Acronym: SPIinChildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: JH2013-2; 2013-003607-19 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-01-27 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Anesthesia
Keywords: Measurement; nosiseption
MeSH Terms: interventions — Levobupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Patients in group receive Ileoinguinal block before the start of surgery, and an injection of plasebo saline after surgery. Injectate is blinded from caregiver.
  Interventions: Drug: Levobupivacaine; Drug: Saline
- Control group (Placebo Comparator): Patients receive a plasebo saline injetion at the site of ileoinguinal block prior to surgery and an injectio with local anesthetics after surgery. The treatment group is blinded for caregiver.
  Interventions: Drug: Levobupivacaine; Drug: Saline

INTERVENTIONS:
Drug: Levobupivacaine
Drug: Saline

SUMMARY:
Surgical Pleth index is a novel device aimed for measurement of intraoperative nosiseption. It has not been tested on small children. The aim of this study is to measure, whether there is a difference in nosiception measured by SPI in a group receiving local anesthetics prior to operation compared to group receiving plasebo.

ELIGIBILITY:
Inclusion Criteria:

* age 0-2 years
* Elective surgery planned for inguinal hernia, or testicle retention
* Written informed consent from parent received
* ASA I-III

Exclusion Criteria:

* Exstrasystolias, known cardiac problem, medication affecting rhytm, allergy to drugs used

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Surgical Pleth Index (SPI) at the time of start of surgery | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Jarkko Harju, MD, Principal Investigator — Tampere University Hospital; Arvi Yli-Hankala, Prof, MD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Harju J, Kalliomaki ML, Leppikangas H, Kiviharju M, Yli-Hankala A. Surgical pleth index in children younger than 24 months of age: a randomized double-blinded trial. Br J Anaesth. 2016 Sep;117(3):358-64. doi: 10.1093/bja/aew215. PMID 27543530